CLINICAL TRIAL: NCT02214524
Title: Comparison of Active Warming System and Conventional Passive Warming Care in Reducing Intraoperative Blood Loss for Patients Undergoing Major Surgery
Brief Title: Comparison of Active and Passive Perioperative Warming Techniques in Reducing Intraoperative Blood Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: 3M (Industry)
Responsible Party: Principal Investigator, Jie YI, Vice director, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MDI0092
Record Dates: First submitted 2014-08-08; First posted 2014-08-12 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Hypothermia; Blood Loss,; Blood Coagulation Disorders
Keywords: perioperative hypothermia; Tympanic temperature; Blood loss; Blood Coagulation Disorders; Major surgery
MeSH Terms: conditions — Hypothermia; Hemorrhage; Blood Coagulation Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bair hugger forced air warming therapy (Experimental): Use of Bair Hugger forced-air warming system perioperatively to keep patient normothermia
  Interventions: Device: Bair Hugger forced air warming system
- conventional warming care (No Intervention): conventional warming care

INTERVENTIONS:
Device: Bair Hugger forced air warming system — Bair Hugger Model 775 temperature management unit-offers two airflow settings, hose-end temperature sensing, and precise temperature delivery
  Other Names: Bair Hugger 775, 70-2007-6800; Bair Hugger Blanket Model 635 and 300
  Arms: Bair hugger forced air warming therapy

SUMMARY:
This is a randomized, open label, parallel two arm, clinical study, which compare the Bair Hugger forced-air warming blanket and the conventional warming care practice in China on patients undergoing major surgery to determine the impact of maintaining normothermia on intraoperative blood loss, requirement for transfusion of packed red blood cells and the changes of coagulation function.

DETAILED DESCRIPTION:
Each Investigator reviews the most current Instructions for Use for Bair Hugger Forced air Warming System to assess the contraindications, warnings, and precaution sections with respect to risks and benefits for treating potential patients.

60 patients will be enrolled preliminary in this clinical trial. Equal size of 30 patients were allocated randomly into interventional or control group.

Randomization will be performed after the patient has met all eligibility criteria, including the general inclusion or exclusion and the patient or legally authorized representative has signed an informed consent form prior to any study related procedure.

Prior to induction, patients in the interventional group were provided 15 to 30 minutes forced air warming using the Bair Hugger warming unit, either in the pre-anesthesia area or OR,which may add to the total heat content of the body helping to reduce the effects of redistribution temperature drop for procedures using a temperature management strategy. The Bair Hugger warming unit is placed on its highest temperature setting and will be adjusted by the investigator depending on temperature monitoring. Temperature will be measured in both groups by either Spot-On sensor and tympanic membrane thermometer.

Statistical analysis will be performed after the data of 30 cases (both groups) were available and the sample size will be re-estimated based on preliminary data analysis. Continuous variables will be summarized with mean, median, standard deviation, minimum and maximum, as applicable. Categorical variables will be summarized with frequency and percentage. Student t test will be used to compare means for continuous variables. A Chi square test or a Fisher's exact test will be used to compare proportions for categorical variables. Multiple regression will be performed to assess the risk ratios of patients developing hypothermia and will be expressed as an risk ratio along with a 95% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients≥18 years old
* Preoperative core temperature between 36.0 and 37.5°C
* American Society of Anaesthesiologists（ASA） Physical Status Classification System I-III
* No transdermal meds on the target site
* Elective major surgeries included but not limited:

  * Hip replacement
  * Thoracic surgery (lobectomy and esophagectomy) or abdominal surgery

Exclusion Criteria:

* Less than 18 years old
* Uncontrolled insulin-dependent diabetes mellitus (preoperative glucose >250 mg/dL)
* A preoperative temperature above 37.5°C or less than 36°C
* Hyperthyroidism and hypothyroidism
* Raynaud disease
* History of infection and fever within 4 weeks before surgery
* Use of steroid or immunosuppressant within 4 weeks before surgery
* History of bleeding disorders
* Clinically significant laboratory abnormalities
* Hgb ≤ 10.0 g/L
* Platelets ≤ 100,000 / mL
* WBC（white blood cell ） <3000/dL
* Fibrinogen<200 mg/dL
* Thromboplastin time>40s
* Prothrombin time
* international normalized ratio(INR）<70%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-08; Primary Completion 2014-11 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Core Temperature and blood loss | intraoperative
  Monitor the changes of core temperature for whole perioperative period and the amount of blood loss were recorded

SECONDARY OUTCOMES:
Length of Stay in PACU | 90 days after Hip replacement surgery and 30 days after other surgerys
Length of Stay in Hospital | 90 days after Hip replacement surgery and 30 days after other surgerys
Length of Stay in ICU | 90 days after Hip replacement surgery and 30 days after other surgerys
Surgical Site Infection（SSI） | 90 days after Hip replacement surgery and 30 days after other surgerys
coagulation function | perioperative period
  take blood sample to detect the coagulation function,including Prothrombin time,Active Partial Thromboplastin Time,International normalized Ratio,Thromboelastography,Hemoglobin,ect.

CONTACTS AND LOCATIONS:
Overall Officials: Yugung Huang Huang, doctoral, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Yi J, Liang H, Song R, Xia H, Huang Y. Maintaining intraoperative normothermia reduces blood loss in patients undergoing major operations: a pilot randomized controlled clinical trial. BMC Anesthesiol. 2018 Sep 8;18(1):126. doi: 10.1186/s12871-018-0582-9. PMID 30193571